CLINICAL TRIAL: NCT07363603
Title: An Open-Label, Non-Randomized Study to Evaluate the Efficacy and Safety of ASO-GNAO1 (Tianasen) in Patients With GNAO1-Encephalopathy With Epilepsy and Movement Disorders Following Repeated Intrathecal Dose Escalation.
Brief Title: Tianasen (ASO-GNAO1) for GNAO1-Encephalopathy With Epilepsy and Movement Disorders.
Acronym: ASO-GNAO1
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pirogov Russian National Research Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASO-GNAO1
Record Dates: First submitted 2025-09-29; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-09

CONDITIONS: GNAO1; Epilepsy; Hyperkinesis
Keywords: GNAO1; Epilepsy; hyperkinesis
MeSH Terms: conditions — Epilepsy; Hyperkinesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GNAO1 c.607G>A carriers (Experimental): Patients enrolled based on the screening results will receive intrathecal administration of the ASO drug Tianasen, starting with a minimum initial dose of 0.3 mg/kg. The drug dose will be escalated every 2 weeks until the expected therapeutic dose of 1.2 mg/kg is reached. With good tolerability, the dose may be further increased to 1.5 mg/kg.
  Upon reaching the final dose level, an interim analysis of the results from the dose escalation period (including PK, efficacy, and safety assessments) will be conducted. Based on the results of this analysis, a decision will be made regarding the continuation of the study using the achieved dose.
  The study may be terminated prematurely if the risk-benefit ratio is deemed unfavorable.
  Interventions: Biological: Antisense oligonucleotide treatment (ASO)

INTERVENTIONS:
Biological: Antisense oligonucleotide treatment (ASO) — Intrathecal escalating doses from 0.3 mg/kg to 1.5 mg/kg (single administration per dose level)
  Other Names: Tianasen

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety of the investigational drug ASO-GNAO1 (Tianasen) in pediatric patients with c.607G>A mutation in the GNAO1 gene associated with epilepsy and neurodevelopmental disorder. The main questions it aims to answer are:

1. Does intrathecal administration of ASO-GNAO1 slow or halt the progression of motor and cognitive symptoms?
2. Is ASO-GNAO1 safe and well-tolerated in this patient population?
3. What is the appropriate therapeutic dose?

This is an open-label study without a placebo control group due to the rare and severe nature of the disease. All participants will receive the active drug.

Participants will:

Receive escalating doses of ASO-GNAO1 via intrathecal injection over a 12-month period.

Undergo frequent neurological assessments, biomarker testing, and safety monitoring.

DETAILED DESCRIPTION:
The variant c.607G>A in the GNAO1 gene is a gain-of-function (GOF) mutation associated with epilepsy and neurodevelopmental disorder.

ASO-GNAO1 (Tianasen) is an investigational antisense oligonucleotide (ASO) therapy designed for the treatment of GNAO1-encephalopathy. Its mechanism of action is allele-specific suppression of the mutant GNAO1 protein expression at the mRNA level. The compound mediates the degradation of mutant mRNA or inhibits its translation, thereby halting the synthesis of the pathogenic protein implicated in disease progression. This targeted suppression is anticipated to mitigate neurodegenerative processes and facilitate partial or complete restoration of neuronal function.

The drug candidate was identified through a screening platform analogous to that used for the development of Milasen, an FDA-authorized personalized ASO therapy for Batten disease. In vitro studies have demonstrated that ASO-GNAO1 (Tianasen) achieves approximately 85% suppression of the mutant GNAO1 allele activity (c.607G>A mutation) while showing no significant effect on the wild-type allele, confirming its allele-specificity.

Background and Rationale. GNAO1 encephalopathy is a severe, debilitating monogenic neurodevelopmental disorder of childhood onset, characterized by progressive motor dysfunction and drug-resistant epilepsy and hyperkinesis. Currently, there are no approved disease-modifying therapies, and management is limited to palliative and symptomatic care. The disease course is progressive, leading to severe developmental delay, profound disability, and premature mortality.

The rationale for this first-in-human study is to evaluate the potential of ASO-GNAO1 (Tianasen) to alter the natural history of the disease in a population with no alternative effective treatment options.

Study Design and Preclinical Rationale. This study constitutes the first human administration of ASO-GNAO1 (Tianasen). It is initiated as an investigational personalized therapeutic development effort for children with a rare monogenic mutation.

The preclinical toxicology program supporting this trial included single- and repeat-dose toxicity studies in rats. Doses were administered at three levels (0.2 mg/kg, 0.5 mg/kg, and 1.0 mg/kg) via intrathecal bolus injection five times over a 12-week period. The maximum observation period in the repeat-dose toxicity study was 141 days (20 weeks). The established No Observed Adverse Effect Level (NOAEL) and the overall design of the abbreviated preclinical package are consistent with the regulatory precedent set by other personalized ASOs, such as Milasen, which was authorized for a single-patient Investigational New Drug (IND) application.

Rationale for Dose Selection. The starting dose and escalation regimen for this study are based on an integrated analysis of the preclinical toxicology data, including the determination of the NOAEL and the estimated maximum tolerated dose. Further justification is derived from the known pharmacokinetic and pharmacodynamic profiles of structurally and mechanistically similar ASO compounds approved for intrathecal administration in neurological diseases, notably nusinersen and the personalized therapy milasen. Dosing is designed to remain within the established safety margins while targeting concentrations anticipated to be therapeutic based on preclinical efficacy models

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent: Written informed consent from the parent(s) or legal guardian(s) of the patient and the child's assent (where applicable based on age and cognitive ability), obtained prior to the initiation of any study-related procedures.
* Age: Male or female children aged 1 year and older (≥1 year) until 14 years at the time of informed consent signing.
* Diagnosis: A confirmed a c.607G>A variant in of GNAO1 gene based on genetic testing, and a clinical presentation that includes both epilepsy and movement disorders.
* Treatment Resistance:

  * For seizures: Documented resistance to antiseizure medications prior to screening, defined as the persistence of seizures despite adequate trials of at least two appropriately dosed antiseizure medications.
  * For non-epileptic hyperkinesias/dystonia: Documented resistance to anti-hyperkinetic medications prior to screening, defined as the persistence of debilitating hyperkinesias or dystonic attacks despite adequate trials of at least two appropriately dosed anti-hyperkinetic medications.
* Contraception (for females of reproductive potential): For post- menarche female adolescents, a negative serum or urine pregnancy test at screening and agreement to use highly effective methods of contraception (e.g., hormonal implants, combined oral contraceptives, intrauterine device) throughout the study participation period.

Exclusion Criteria:

* Unacceptable Risk: Any concurrent severe medical, neurological, or psychiatric condition, or any other significant circumstance (e.g., unstable clinical status) that, in the judgment of the Investigator, could significantly increase the risk associated with study participation or the administration of the investigational product, or could interfere with the interpretation of study results.
* Impossibility of Intervention: Any anatomical abnormality, coagulation disorder, active infection, or other condition that constitutes a contraindication to or precludes the safe performance of repeated lumbar punctures for intrathecal administration of the study drug.
* Pregnancy or Lactation: Pregnancy, lactation, or intention to become pregnant during the study period.
* Concurrent Experimental Therapy: Receipt of any other investigational drug, device, or biological product within 1 month prior to screening or within a period of at least 5 half-lives of that product (whichever is longer).
* Protocol Compliance: Any other disease, condition, or behavioral factor that, in the opinion of the Investigator, could compromise the patient's safety, preclude adherence to the protocol schedule, or interfere with the study conduct and endpoint assessments. Age: 14 years and older

Ages: 1 Year to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Estimated)
Dates: Start 2025-09-09 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in monthly seizure frequency | Baseline to Week 50
  Change from Baseline in the number of seizure episodes per month. Unit of Measure: seizures per month
Change in total monthly duration of seizures | Baseline to Week 50
  Change from Baseline in the total duration of seizure episodes per month.
  Unit of Measure: minutes per month
Change in frequency of non-epileptic hyperkinetic and dystonic episodes | Baseline to Week 50
  Change in frequency of non-epileptic hyperkinetic and dystonic episodes
  Unit: episodes per month
Change in duration of non-epileptic hyperkinetic and dystonic episodes | Baseline to Week 50
  Change in duration of non-epileptic hyperkinetic and dystonic episodes
  Unit: minutes per month

SECONDARY OUTCOMES:
Change in epileptiform activity index on EEG | Baseline, Week 46
  Change from Baseline in the quantitative EEG epileptiform activity index.
  Unit of Measure: percentage of recording time with epileptiform activity
  Range of Measure: 0-100%, higher value = worse
Change in Barry-Albright Dystonia Scale score | Baseline, Week 46
  Change in Barry-Albright Dystonia Scale score Unit: score (0-160), higher scores indicate worse dystonia
Change in concomitant medication dosages | Baseline, Week 46
  Change in total daily medication dose
  Unit: mg/kg/day
Change in Gross Motor Function Measure-88 total score | Baseline, Week 46
  Change in Gross Motor Function Measure-88 total score
  Unit: score (0-100), higher scores indicate better function
Change in Denver Developmental Screening Test developmental age | baseline and week 46
  Change in Denver Developmental Screening Test developmental age
  Unit: developmental age in months
Change in Leiter-3 nonverbal IQ score | Baseline and week 46
  Change in Leiter-3 nonverbal IQ score.
  Unit: IQ score (standard score 30-170)

CONTACTS AND LOCATIONS:
Overall Officials: Elena D Belousova, Prof, Principal Investigator — Pirogov Russian National Research Medical University
Locations (1):
- Veltischev Research and Clinical Institute for Pediatrics and Pediatric Surgery of the Pirogov Russian National Research Medical University, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication are to be shared
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: immediately after the publication of the final article in a peer-reviewed journal and ending 3 years after the publication of results
Access Criteria: Access to de-identified IPD will be granted to researchers affiliated with academic or scientific research institutions, as well as to representatives of pharmaceutical companies, provided that the request is approved by the study's Scientific Steering Committee.
  Applicants must submit a formal request to bv@mda-cro.com. The request must include a detailed description of the research question, analysis plan, required set of variables, and timeline. The Committee's decision will be based on the scientific merit of the proposal, the ethical nature of the objectives, and data availability.
  Approved applicants will be required to sign a Data Transfer Agreement (DTA), which obligates them to use the data solely for the stated purpose, not to attempt to re-identify participants, to ensure data security, and to acknowledge the original source in any publications. The analysis must be conducted in accordance with the pre-approved statistical plan.